CLINICAL TRIAL: NCT05431868
Title: Presbyopia-correcting Performance and Subjective Outcomes of a Trifocal Intraocular Lens in Eyes With Different Axial Lengths: a Prospective Cohort Study
Brief Title: Objective and Subjective Outcomes of a Trifocal IOL in Eyes With Different AL
Status: Completed | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Trifocal&AL
Record Dates: First submitted 2022-06-20; First posted 2022-06-24 (Actual); Last update posted 2022-06-24 (Actual); Status verified 2022-06

CONDITIONS: Cataract; Presbyopia; Lenses, Intraocular; Myopia; Satisfaction
Keywords: Cataract; Presbyopia; Intraocular Lens; Axial Length; Satisfaction
MeSH Terms: conditions — Cataract; Presbyopia; Myopia; Personal Satisfaction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- the short AL group: Eyes with AL less than 22.50 mm were devided into the short AL group.
  Interventions: Other: AT LISA tri 839MP (Carl Zeiss Meditec AG)
- the control group: Eyes with AL between 22.50 to 25.50 mm were devided into the control group.
  Interventions: Other: AT LISA tri 839MP (Carl Zeiss Meditec AG)
- the long AL group: Eyes with AL more than 25.50 mm were devided into the long AL group.
  Interventions: Other: AT LISA tri 839MP (Carl Zeiss Meditec AG)

INTERVENTIONS:
Other: AT LISA tri 839MP (Carl Zeiss Meditec AG) — This prospective cohort study collected data of patients who underwent bilateral or unilateral cataract surgery with the AT LISA tri 839MP implantation.

SUMMARY:
This prospective cohort study enrolled patients with implantation of a trifocal IOL. Only one eye of each patient was enrolled. Eyes were devided into three groups according the axial length (AL), including the short AL group, the control group and the long AL group. Manifest refraction, uncorrected and distance-corrected visual acuity at different distances, contrast sensitivity, aberrations and IOL decentration were measured three months after surgery. Spectacle independence, adverse photic phenomena, overall satisfaction and life quality were assessed with a questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria were patients older than 40 years with significant bilateral or unilateral cataract seeking spectacle independence, with the AL between 21.00 to 30.00 mm, the prediction of postoperative corneal astigmatism less than 1.0 diopters (D), the angle kappa less than 0.50 mm, the corneal spherical aberration less than 0.5 μm and the corneal higher order aberration less than 0.5 μm.

Exclusion Criteria:

* Exclusion criteria were eyes with serious intraoperative complications, irregular corneal astigmatism, corneal scarring, uveitis, glaucoma, pseudoexfoliation syndrome, macular degeneration or other retinal impairment, amblyopia or patients having difficulties with examinations or 3 months' follow-up.

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This prospective cohort study collected data of patients who underwent bilateral or unilateral cataract surgery with the AT LISA tri 839MP implantation at the Department of Ophthalmology, Peking University Third Hospital, Beijing, China.
Sampling Method: Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Refractive Outcomes | Three months after surgery.
  Manifest refraction was measured.
Visual Acuity at Different Distances | Three months after surgery.
  Uncorrected and corrected distance (5 m) visual acuity (UDVA, CDVA), uncorrected and distance-corrected intermediate (80 cm) and near (40 cm) visual acuity (UIVA, DCIVA, UNVA and DCNVA) were measured.
Defocus Curve | Three months after surgery.
  The defocus curve was measured with the additional spherical diopters from +2.00 D to -4.00 D in 0.50 D steps.
Contrast Sensitivity and Aberrations | Three months after surgery.
  Using the OPTEC 6500 Vision Tester (Stereo Optical Co. Inc, Chicago, USA), the contrast sensitivity was conducted under four conditions, including photopic(85 cd/m2), mesopic(3 cd/m2), photopic with glare and mesopic with glare. Besides, there are five spatial frequencies (1.5, 3, 6, 12, and 18 cycles per degree [cpd]) under every condition.
IOL decentration | Three months after surgery.
  OPD Scan-III (NIDEK, Inc.) can automatically recognize and locate the edge of the pupil and measure its position relative to the optic axis. After pupil dilation, the IOL decentration was measured through adjusting the edge of the pupil to the edge of the lens manually.
Subjective Satisfaction | Three months after surgery.
  The subjective satisfaction was assessed by a self-made questionnaire, which evaluated the spectacle independence at different distances, the incidence of several adverse photic phenomena including glare, halo and starburst, and the overall satisfaction.
Life Quality | Three months after surgery.
  The life quality after surgery was assessed by the National Eye Institute Visual Function Questionnaire-25 (NEI VFQ-25) in Chinese.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided